CLINICAL TRIAL: NCT04782557
Title: Endoscopic Ultrasound Guided Hepatic and Portal Vein Aspiration for Circulating Tumor DNA in Patients Suffering From GI Cancers
Brief Title: EUS Guided HVA and PVA for Circulating Tumor DNA in Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHAN SHANNON MELISSA, Assistant professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020.321
Record Dates: First submitted 2021-01-05; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Circulating Tumor Cell; Gastrointestinal Cancer
Keywords: Circulating Tumor Cell; Gastrointestinal Cancer; Endoscopic ultrasound portal vein aspiration
MeSH Terms: conditions — Neoplastic Cells, Circulating; Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EUS-guided PVA and HVA (Experimental): Patient will undergo EUS-guided PVA and HVA
  Interventions: Diagnostic Test: EUS-guided portal vein and hepatic vein aspiration

INTERVENTIONS:
Diagnostic Test: EUS-guided portal vein and hepatic vein aspiration — EUS-guided portal vein and hepatic vein aspiration

SUMMARY:
The discovery of cell-free circulating tumor DNA (crDNA) in blood and the maturation of technologies for ctDNA analysis have presented an attractive opportunity for minimally invasive "liquid biopsy" genomic diagnostics. The investigators plan to perform EUS-guided portal vein and hepatic vein aspiration in GI cancers patients. The aim of the current study is thus to examine the concentration of ctDNA in portal vein (EUS-guided PVA), hepatic vein (EUS-guided HVA) and peripheral blood to understand the first pass effect of the liver with gastrointestinal (GI) cancers, and the possibility of using ctDNA as a marker for preoperative staging, restaging after neoadjuvant chemotherapy, and monitoring for recurrence.

DETAILED DESCRIPTION:
The discovery of cell-free circulating tumor DNA (crDNA) in blood and the maturation of technologies for ctDNA analysis have presented an attractive opportunity for minimally invasive "liquid biopsy" genomic diagnostics. The investigators plan to perform EUS-guided portal vein and hepatic vein aspiration in GI cancers patients. The aim of the current study is thus to examine the concentration of ctDNA in portal vein (EUS-guided PVA), hepatic vein (EUS-guided HVA) and peripheral blood to understand the first pass effect of the liver with gastrointestinal (GI) cancers, and the possibility of using ctDNA as a marker for preoperative staging, restaging after neoadjuvant chemotherapy, and monitoring for recurrence.

ELIGIBILITY:
Inclusion criteria:

1. Age >= 18 years old
2. Newly diagnosed stage II-IV distal gastric cancer, pancreatic cancer or colorectal cancer
3. Undergoing treatment with either:

   1. Surgery
   2. Neoadjuvant chemotherapy
   3. Neoadjuvant chemoirradiation
   4. Palliative chemotherapy/ immunotherapy

      Exclusion criteria:

   <!-- -->

   1. Synchronous cancer of other sites
   2. Cardia, high lesser curve tumors, oesophagogastric junction tumors
   3. Presence of bulky lymph nodes at lesser curve/ coeliac region precluding a clear EUS puncture site to portal vein and hepatic vein
   4. Patients with coagulopathy (international normalized ratio >1.3, partial thromboplastin time greater than twice that of control), platelet count <50,000x103/uL
   5. Patients unwilling to undergo follow-up assessments
   6. Patients with liver cirrhosis, portal hypertension and/ or gastric varices
   7. Patient refusal to participate

      -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Variant allelic fraction (expressed in %) of serum ctDNA from HVB, PVB and peripheral blood | 3 months
  Plasma DNA will be extracted using the QIAamp Circulating Nucleic Acid Kit (Qiagen), and the concentration of the circulating tumor DNA will be reported in variant allelic fraction (expressed in %)

SECONDARY OUTCOMES:
Variant allelic fraction (expressed in %) of Genomic and proteomic analysis of ctDNA | 3 months
  If ctDNA is identified, further genomic and proteomic analysis will be performed. It will be measured in terms variant allelic fraction (expressed in %)
Staging of the GI cancer | 3 months
  The pathological TNM staging of the resected specimen will be recorded.
Recurrence | 5 years
  any recurrence of the tumor will be recorded
Overall survival | 5 years
  overall survival will be recorded
Progression-free survival | 5 years
  progression free survival will be recorded
Technical success rate of EUS-PVA and HVA | 1 day
  The technical success rate of the EUS guided procedure will be recorded. Reasons for failure of the cases will be recorded.
Adverse events of EUS-PVA and HVA | 30 days
  the adverse events of the EUS procedure will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No